CLINICAL TRIAL: NCT01659346
Title: A Prospective Randomized Controlled Trial Comparing Non-selective Beta Blockers Versus EVL for Primary Prophylaxis of Esophageal Variceal Bleeding in Patients With Hepatocellular Carcinoma With Portal Vein Tumour Thrombosis
Brief Title: Non-selective Beta Blockers Versus EVL for Primary Prophylaxis of Esophageal Variceal Bleeding in Patients With Hepatocellular Carcinoma With Portal Vein Tumour Thrombosis.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to high mortality
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-HCC-01
Record Dates: First submitted 2012-08-04; First posted 2012-08-07 (Estimated); Last update posted 2017-11-17 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma With Portal Vein Thrombosis
MeSH Terms: interventions — Carvedilol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Endoscopic Variceal Ligation (Experimental): Endoscopic Variceal Ligation every 3 weeks till eradication
  Interventions: Procedure: Endoscopic Variceal Ligation
- Carvedilol (Active Comparator): Carvedilol 3.125mg BD increased after 1 week to reach 6.25mg BD
  Interventions: Drug: Carvedilol

INTERVENTIONS:
Procedure: Endoscopic Variceal Ligation — Endoscopic Variceal Ligation every 3 weeks till eradication.
  Arms: Endoscopic Variceal Ligation
Drug: Carvedilol — Carvedilol 3.125mg BD increased after 1 week to reach 6.25mg BD
  Arms: Carvedilol

SUMMARY:
Every patient with HCC (Hepato-Cellular Carcinoma) with main portal vein thrombosis will be screened for presence of large esophageal varices and will be randomized between non-selective beta blocker versus primary endoscopic variceal ligation. They will be followed to assess the rate of reduction of index bleed rate as well as survival difference between the groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients of cirrhosis with Hepatocellular carcinoma and portal vein thrombosis
* Presence of large oesophageal varices or small with high risk

Exclusion Criteria:

* Any contra-indication to beta-blockers
* Any Endoscopic Variceal Ligation or Sclerotherapy within last 3 months
* High risk gastric varices
* Any past history of Transhepatic Intrajugular Portosystemic Shunt or surgery for portal hypertension
* Significant cardio or pulmonary co-morbidity
* Any extrahepatic malignancy
* Patients with past history of variceal bleed
* Patients with non-tumor portal vein thrombosis
* Refusal to participate in the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-02; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
First Variceal Bleeding | 1.5 years

SECONDARY OUTCOMES:
Death | 1.5 years
Procedure related complications. | 1.5 years
Reappearance of Esophageal varices in presence of Portal Vein Thrombosis | 1.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Dr Shakti P Choudhury, MD, Principal Investigator — Institute of Liver and Biliary Sciences
Locations (1):
- Institute of Liver and Biliary Sciences, New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: Undecided